CLINICAL TRIAL: NCT06097026
Title: Role of Inhaled Nitric Oxide in Vascular Mechanics and Right Ventricular Function Following Cardiac Surgery
Brief Title: Role of Inhaled Nitric Oxide in Vascular Mechanics and Right Ventricular Function
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fernando Suarez Sipmann (Other)
Collaborators: Air Liquide SA (Industry)
Responsible Party: Sponsor-Investigator, Fernando Suarez Sipmann, MD PhD Intesive Care Medicine, Principal Investigator, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RONNIN- CCV
Record Dates: First submitted 2023-09-26; First posted 2023-10-24 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Collapsed Lung; Hemodynamic Stability
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Nitric Oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard treatment (CONT) (No Intervention): The patient will be managed according to the routine clinical protocol, homogenizing the interventions in both participating centers.
- iNO 20-40 ppm (Experimental): In this arm, inhaled nitric oxide therapy will be initiated at 20 ppm immediately after randomization and after initial data collection. The dose will be reassessed after the first 30 min and may be increased to a maximum of 40 ppm depending on the response observed in ventricular function.
  Interventions: Drug: Nitric Oxide
- iNO 20 - 40 ppm + Lung recruitment (iNO-RM) (Experimental): After 30 min after initiation of nitric oxide therapy following randomization, once patient stability has been confirmed, a brief recruitment maneuver will be performed and the subsequent PEEP level will be individualized according to the best lung compliance. Ventilation will then continue with the standard baseline ventilator settings, but with the PEEP level individually optimized.
  Interventions: Procedure: Alveolar recruitment maneuver; Drug: Nitric Oxide

INTERVENTIONS:
Procedure: Alveolar recruitment maneuver — Progressive pressure increase on the ventilator to recruit collapsed alveoli and improve pulmonary ventilation.
  Other Names: Alveolar recruitment
  Arms: iNO 20 - 40 ppm + Lung recruitment (iNO-RM)
Drug: Nitric Oxide — Administer nitric oxide upon arrival from cardiac surgery and assess cardiac and pulmonary function afterwards.
  Arms: iNO 20 - 40 ppm + Lung recruitment (iNO-RM); iNO 20-40 ppm

SUMMARY:
The aim of this study is to evaluate the role of nitric oxide on pulmonary vasculature and right ventricular function in postoperative cardiac surgery patients.

DETAILED DESCRIPTION:
This study will evaluate modifiable pathophysiological treatments for postoperative pulmonary hypertension and right ventricular dysfunction.

One pharmacological, inhaled nitric oxide, and one non-pharmacological, the OLA strategy combining lung recruitment and stabilization with individually optimized positive end-expiratory pressure (PEEP) and the possible synergistic effects of both interventions on right ventricular performance. Apart from acting specifically on the pathophysiological mechanisms described, the combination of an OLA strategy and iNO may be particularly beneficial, as modification of pulmonary status by OLA may, in theory, enhance the effects of iNO by significantly increasing gas exchange area and thus alveolar ventilation.

A number of closely related physiological variables will also be studied to better characterize the effects of both strategies and their combination. This may help to better establish the indication for iNO in cardiac surgery patients and improve our understanding of mechanisms that are also present in ARDS patients, albeit on a different scale.

This is a prospective randomized controlled physiological prospective study to be performed in two hospitals. The intervention period is limited to the first 2 -3 hours postoperatively. A total of 54 patients will be recruited.

ELIGIBILITY:
* Age > 18 years
* Under controlled mechanical ventilation in passive conditions
* Presence of postoperative lung collapse (confirmed by pulmonary echocardiography and Air test)
* Preoperative left ventricular ejection fraction (LVEF) ≥ 30%.
* Absence of hypovolemia: absence of "kissing" ventricles and/or collapsibility index of the superior vena cava < 20%.
* Stable spontaneous heart rhythm
* Postoperative hemodynamic stability:
* Mean arterial pressure (MAP) ≥ 60 mmHg
* Central venous pressure (CVP) ≥ 10 mmHg
* Heart rate (HR) ≤ 100 bpm without tachyarrhythmias
* Lactic acid ≤ 3 mmol/L
* Single vasopressor treatment
* Norepinephrine dose ≤ 0.2 μg/kg/min, without an increase ≥ 15% in the last 30 -minutes.

Obtained informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Right ventricular cardiac function specifically those directly related to the estimation ofright ventricular-vascular coupling | A first TTE baseline measurement (T1) will be taken after arrival in the ICU after cardiac surgery, then another measurement will be taken 30 minutes after the first intervention (at iNO) (T2), and a new measurement will be taken 30 minutes later (T3).
  The parameters will be evaluated by TEE. Right ventricular function parameters will be assessed by the ratio of right ventricular end-diastolic to left ventricular end-diastolic diameters, right ventricular shortening fraction, tricuspid annular plane systolic excursion (TAPSE), myocardial performance index (MPI). estimation of systolic pulmonary artery pressure (PAPs), estimation of pulmonary vascular resistance by Doppler, Right ventricular outflow tract notch pattern, right ventricular outflow tract acceleration time (RVOT-AT).

SECONDARY OUTCOMES:
Electrical impedance tomography (EIT) derived variables | A first baseline measurement (T1) will be taken after arrival at the ICU after cardiac surgery, then another measurement will be taken 30 minutes after the first intervention (in iNO) (T2), and a new measurement will be taken 30 minutes later (T3).
  With electrical impedance tomography (EIT), investigators will analyze the regional distribution of lung ventilation and percussion, the relative distribution of ventilation and percussion in predefined regions of interest, changes in lung aeration (end-expiratory lung volume difference) and pulmonary artery pulsatility.

CONTACTS AND LOCATIONS:
Locations (1):
- Fernando Suárez Sipmann, Madrid, Spain

DOCUMENTS (1):
  • Study Protocol (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT06097026/Prot_000.pdf